CLINICAL TRIAL: NCT03967808
Title: French Renal Epidemiology and Information Network (REIN) Registry in Lorraine
Brief Title: French Renal Epidemiology and Information Network (REIN) Registry
Acronym: REIN-LOR
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Principal Investigator, Carole AYAV, Doctor, Central Hospital, Nancy, France
Other Study IDs: REIN-01
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: End-stage Renal Disease
Keywords: Registry; Renal replacement therapy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Renal Epidemiology and Information Network (REIN) Registry was created in 2002 (after study pilot in 2001) to contribute to the development and evaluation of health strategies aiming at improving prevention and management of end-stage renal disease, and promoting clinical and epidemiological research in this field. It relies on a network of nephrologists, epidemiologists, patients and public health representatives, coordinated regionally and nationally.

DETAILED DESCRIPTION:
The REIN registry is intended to include all end stage renal disease patients on renal replacement therapy (RRT) - either dialysis or transplantation - living in Lorraine area.

New (incident) patients are reported from the first day of RRT. Patients with a diagnosis of acute renal failure are excluded, i.e. those who recover all or some renal function within 45 days or are considered as such by experts when they die before 45 days. Patients with pre-emptive grafts and those living with a functioning graft are identified from the transplant database.

A set of basic items, including fixed and annually updateable items, was defined for all dialysis patients. Five types of events are reported to the registry on occurrence from the first day of any treatment: (1) renal transplantation, (2) changes in dialysis setting, (3) changes in type of dialysis, (4) transient recovery of renal function and (5) death.

The participation rate of centres in Lorraine is 100%. A clinical research assistant visits every dialysis centre to verify the completeness of patient and event registration, by comparing reports to the registry with centre administration files.

The REIN guide defines all items to be recorded, includes coding instructions, and serves as a standard for all participating regions.

REIN consists of a partnership network and professionals whose Biomedicine Agency is the institutional support. The National level consists of a national coordination, a steering group and a scientific board. Regional level includes a Regional Steering Group led by nephrologist and epidemiological coordinators and an epidemiological unit.

ELIGIBILITY:
Inclusion Criteria:

* All patients with end stage renal disease on renal replacement therapy

Exclusion Criteria:

* Patients with acute renal failure ( i.e. those who recover all or some renal function within 45 days or are considered as such by experts when they die before 45 days)
* Patient's refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All new patients reaching end-stage chronic renal failure and requiring support by a renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2001-01 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of end stage renal disease in Renal Replacement therapy | One year
  New (incident) patients are reported from the first day of Renal Replacement Therapy - either dialysis or renal transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Laurain, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Nephrology unit, University hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided
Open to partnership

REFERENCES:
- [Background] Lassalle M, Ayav C, Frimat L, Jacquelinet C, Couchoud C; Au Nom du Registre REIN. The essential of 2012 results from the French Renal Epidemiology and Information Network (REIN) ESRD registry. Nephrol Ther. 2015 Apr;11(2):78-87. doi: 10.1016/j.nephro.2014.08.002. Epub 2014 Nov 1. PMID 25457107
- [Background] Couchoud C, Stengel B, Landais P, Aldigier JC, de Cornelissen F, Dabot C, Maheut H, Joyeux V, Kessler M, Labeeuw M, Isnard H, Jacquelinet C. The renal epidemiology and information network (REIN): a new registry for end-stage renal disease in France. Nephrol Dial Transplant. 2006 Feb;21(2):411-8. doi: 10.1093/ndt/gfi198. Epub 2005 Oct 18. PMID 16234286